CLINICAL TRIAL: NCT02110732
Title: Lactobacillus Rhamnosus GG in the Middle Ear and Adenoid Tonsil After Randomized, Double-blind, Placebo-controlled Oral Administration
Brief Title: Lactobacillus Rhamnosus GG in the Middle Ear and Adenoid Tonsil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Finnish Institute for Health and Welfare (Other Government)
Responsible Party: Principal Investigator, Anne pitkäranta, Professor/Chief Physician at Hospital District of Helsinki and Uusimaa, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: HelsinkiUCH
Record Dates: First submitted 2014-03-11; First posted 2014-04-10 (Estimated); Results first posted 2021-05-11 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Upper Respiratory Infection; Acute Otitis Media
MeSH Terms: conditions — Respiratory Tract Infections; Otitis Media

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lactobacillus rhamnosus GG (Active Comparator): Lactobacillus rhamnosus GG 8-9 x 10 -9 pmy 2x2 for 3 weeks
  Interventions: Dietary Supplement: Lactobacillus rhamnosus GG
- Crystalline cellulose (Placebo Comparator): Crystalline cellulose
  Interventions: Dietary Supplement: Lactobacillus rhamnosus GG

INTERVENTIONS:
Dietary Supplement: Lactobacillus rhamnosus GG

SUMMARY:
The purpose of this study is to evaluate the effect of oral administration of probiotic Lactobacillus rhamnosus GG in middle ear and adenoid tonsil.

ELIGIBILITY:
Inclusion Criteria:

* recurrent otitis media
* secretory otitis media
* chronic rhinitis
* recurrent sinusitis

Exclusion Criteria:

* significant illness

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2011-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to share IPD.

REFERENCES:
- [Derived] Tapiovaara L, Lehtoranta L, Swanljung E, Makivuokko H, Laakso S, Roivainen M, Korpela R, Pitkaranta A. Lactobacillus rhamnosus GG in the middle ear after randomized, double-blind, placebo-controlled oral administration. Int J Pediatr Otorhinolaryngol. 2014 Oct;78(10):1637-41. doi: 10.1016/j.ijporl.2014.07.011. Epub 2014 Jul 18. PMID 25085073

RESULTS

PARTICIPANT FLOW:
Groups:
- Lactobacillus Rhamnosus GG: Lactobacillus rhamnosus GG 8-9 x 10 -9 pmy 2x2 for 3 weeks
  Lactobacillus rhamnosus GG
- Crystalline Cellulose: Crystalline cellulose
  Lactobacillus rhamnosus GG
Period: Overall Study
Arm/Group | Lactobacillus Rhamnosus GG | Crystalline Cellulose
Started | 20 | 20
Completed | 14 | 17
Not Completed | 6 | 3
Not completed — Physician Decision | 5 | 2
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lactobacillus Rhamnosus GG | Crystalline Cellulose | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 20 | 40
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 12 | 11 | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Finland | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Lactobacillus Rhamnosus GG in Middle Ear Effusion and Adenoid Tonsil
Description: Presence of Lactobacillus rhamnosus GG in middle ear effusion of children having tympanostomy after oral administration of L. GG.
Time Frame: After 3 weeks of oral consumption
Population: Number of participants with tympanostomy
Measure: Count of Units; unit: Samples
Units Other Than Participants: Samples
Arm/Group | Lactobacillus Rhamnosus GG | Crystalline Cellulose
Number analyzed (Participants) | 10 | 3
Number analyzed (Samples) | 19 | 6
Samples | 4 | 1
Statistical Analysis 1: Comparison: Lactobacillus Rhamnosus GG vs Crystalline Cellulose; Test type: Other; p = 0.05, Fisher Exact

2. Secondary Outcome: Presence of Bacterial Pathogens in Middle Ear Effusion Samples
Description: Association of Lactobacillus rhamnosus GG with occurrence of bacterial pathogens in the middle ear.
Time Frame: After 3 weeks of oral consumption
Population: Number of participants with tympanostomy
Measure: Count of Units; unit: Samples
Units Other Than Participants: Samples
Arm/Group | Lactobacillus Rhamnosus GG | Crystalline Cellulose
Number analyzed (Participants) | 10 | 3
Number analyzed (Samples) | 19 | 6
Samples | 12 | 3
Statistical Analysis 1: Comparison: Lactobacillus Rhamnosus GG vs Crystalline Cellulose; Test type: Superiority; p < 0.05, Chi-squared; Categorical variables were analyzed with Chi-square test or Fisher's exact test. Comparisons between groups were by Levene's test for equality of variances. A P-level <0.05 was considered statistically significant. Data were analyzed with SPSS v.19 and NCSS

3. Secondary Outcome: Presence of Rhinovirus and Enterovirus in Middle Ear Effusion Samples
Description: Association of Lactobacillus rhamnosus GG with occurrence of viral pathogens in the middle ear.
Time Frame: After 3 weeks of oral consumption
Population: Number of participants with tympanostomy
Measure: Count of Units; unit: Samples
Units Other Than Participants: Samples
Arm/Group | Lactobacillus Rhamnosus GG | Crystalline Cellulose
Number analyzed (Participants) | 10 | 3
Number analyzed (Samples) | 19 | 6
Samples | 11 | 1
Statistical Analysis 1: Comparison: Lactobacillus Rhamnosus GG vs Crystalline Cellulose; Test type: Superiority; p < 0.05, Chi-squared

ADVERSE EVENTS:
Arm/Group | Lactobacillus Rhamnosus GG | Crystalline Cellulose
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No